CLINICAL TRIAL: NCT01928082
Title: The Effects of Estrogen Replacement Therapy in Postmenopausal Women With Hypercalciuria and Low Bone Mass
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The fellow conducting the recruitment and screening left the institution
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0062
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-10

CONDITIONS: Hypercalciuria; Hypercalciuria, Familial Idiopathic; Osteopenia; Osteoporosis
Keywords: Hypercalciuria, Familial Idiopathic; Hypercalciuria; Osteopenia; Osteoporosis; Postmenopausal women
MeSH Terms: conditions — Hypercalciuria; Hypercalciuria, Absorptive, 2; Bone Diseases, Metabolic; Osteoporosis | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transdermal estradiol (Experimental): Transdermal estradiol 0.05 mg/day for 4 weeks, followed by 0.10 mg/day for 4 weeks
  Interventions: Drug: Transdermal estradiol

INTERVENTIONS:
Drug: Transdermal estradiol — 4 weeks of Vivelle-Dot 0.05 mg/day followed by 4 weeks of Vivelle-Dot 0.10 mg/day
  Other Names: Vivelle-Dot 0.05 mg/day; Vivelle-Dot 0.10 mg/day

SUMMARY:
The purpose of this study is to assess if estrogen replacement normalizes urinary calcium excretion in postmenopausal women with hypercalciuria and low bone mass and to assess for differences in response to estrogen replacement in women with familial hypercalciuria compared to nonfamilial hypercalciuria.

DETAILED DESCRIPTION:
Subjects will primarily be recruited from the subjects of protocol 12-1421. Subjects may also be identified through chart review of patients seen by Dr. Favus in the Bone Clinic at the University of Chicago. These subjects will be mailed a letter describing the study and a request to contact us if they are willing to participate in the study.

We plan to enroll 20 subjects to obtain complete data on 16 subjects. We aim to have 10 subjects who will have confirmed familial idiopathic hypercalciuria (IH) and 10 subjects who will have no family history of hypercalciuria.

Subjects will be brought into the Clinical Research Center at the University of Chicago where blood samples will be collected by phlebotomy to obtain the following screening tests: complete metabolic panel; including calcium, phosphate, magnesium, creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and albumin; parathyroid hormone, 25-hydroxyvitamin D, follicle stimulating hormone (FSH), and estradiol. A twenty-four hour urine collection starting with second void of the day will be collected for calcium, phosphate, magnesium, citrate, oxalate, sodium, ammonia, sulfate, and creatinine. Subjects on diuretics will be screened after a 2 week washout period, provided this can be discontinued safely. If subjects have participated in study protocol number 12-1421, these screening tests do not have to be repeated and the results from protocol number 12-1421 will be used to determine eligibility.

Screening subjects who meet inclusion criteria can proceed to the observational study. Screening subjects who are vitamin D depleted (serum 25-hydroxyvitamin D less than 35 ng/mL) may be rescreened after repletion of vitamin D.

A letter describing the study aims, protocols, and risks and benefits will be sent to their primary care physicians and gynecologists. Upon completion of the study, a summary letter will be sent as well.

Prior to the baseline visit a twenty-four hour urine collection starting with the second void of the day will be collected for calcium, phosphate, magnesium, citrate, oxalate, sodium, ammonia, sulfate, and creatinine. Subjects on diuretics will require a 2 week washout period, provided this can be discontinued safely. During the baseline visit a medical history will be taken and a physical exam will be performed. Venous blood will be collected for 1,25-dihydroxyvitamin D3, osteocalcin, bone-specific alkaline phosphatase, C-telopeptides of type 1 collagen (CTX), procollagen type 1 N-terminal propeptide (P1NP), bone morphogenetic protein 2 (BMP-2), and sclerostin. If the subject has had these blood tests performed in the preceding four months for protocol 12-1421, the blood tests will not be repeated. 18F sodium fluoride PET/CT bone scan will be performed. The protocol for the radionuclide imaging is attached.

All subjects will be started on transdermal 17-beta-estradiol 0.05 mg/d, which is equivalent to the standard dose of conjugated estrogen dose of 0.625 mg, for 4 weeks and increased to 0.1 mg for subsequent 4 weeks. Given the short duration of this study, progesterone will not be provided, as 8 weeks is not of sufficient duration to significantly increase the risk of endometrial cancer (Strom, Schinnar et al. 2006).

For the entire study, diuretics will be discontinued if it has been deemed safe to do so by the principle investigator or prescribing physician. Throughout the study, subject will maintain 900-1200 mg of dietary calcium daily. To monitor dietary calcium intake, a 5 day diet diary will be kept from Sunday to Thursday of the fourth week of each medication dose. Compliance of the study medication will be assessed by estrogen patch counts.

The following blood tests will be repeated 4 and 8 weeks after starting estradiol patch: complete metabolic panel (including calcium, phosphate, potassium, bicarbonate, chloride, magnesium, creatinine, and albumin), 25-hydroxyvitamin D, 1,25-dihydroxyvitamin D3, parathyroid hormone, estradiol, osteocalcin, bone-specific alkaline phosphatase, C-telopeptides of type 1 collagen (CTX), procollagen type 1 N-terminal propeptide (P1NP), bone morphogenetic protein 2 (BMP-2), and sclerostin. In addition, 4 and 8 weeks after starting estradiol patch, 24 hour urine collection will be performed for calcium, phosphate, magnesium, citrate, oxalate, sodium, ammonia, sulfate, and creatinine.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Diagnosis of hypercalciuria
* Diagnosis of low bone mass
* Vitamin D replete (serum 25-hydroxyvitamin D level >35 ng/mL)

Exclusion Criteria:

* Secondary causes of hypercalciuria (primary hyperparathyroidism, sarcoidosis, vitamin D excess, malignant neoplasm, and renal tubular acidosis)
* Other metabolic bone disease (primary hyperparathyroidism, hyperthyroidism, hypercortisolemia, severe gastrointestinal disorders, liver cirrhosis, renal failure (Cr >1.5), active malignancy including multiple myeloma, rheumatological diseases, and Paget's disease of bone)
* Use of medications affecting bone and calcium metabolism (corticosteroids in the previous 3 months, suppressive dose of thyroid hormone, calcium channel blockers, anti-convulsants, aromatase inhibitors, thiazolidinediones, and cyclosporine A)
* History of coronary artery disease
* Breast cancer or suspected estrogen-dependent neoplasia
* Previous venous thromboembolic event
* Stroke
* Active liver disease
* Tobacco use within the past 6 months
* Negative colonoscopy within the previous 10 years or sigmoidoscopy within the previous 5 years
* Negative mammogram within the previous 2 years
* Negative Pap smear within the previous 3 years in women < or = 65 years old with an intact cervix
* No vaginal bleeding within the prior 5 months.
* Age > or = 70
* > or = 20 years since last menstrual period or use of hormone replacement therapy

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray J Favus, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Cerda Gabaroi D, Peris P, Monegal A, Albaladejo C, Martinez MA, Muxi A, Martinez de Osaba MJ, Suris X, Guanabens N. Search for hidden secondary causes in postmenopausal women with osteoporosis. Menopause. 2010 Jan-Feb;17(1):135-9. doi: 10.1097/gme.0b013e3181ade8e5. PMID 19593233
- [Background] Christiansen C, Riis BJ, Rodbro P. Prediction of rapid bone loss in postmenopausal women. Lancet. 1987 May 16;1(8542):1105-8. doi: 10.1016/s0140-6736(87)91671-0. PMID 2883442
- [Background] Deutschmann HA, Weger M, Weger W, Kotanko P, Deutschmann MJ, Skrabal F. Search for occult secondary osteoporosis: impact of identified possible risk factors on bone mineral density. J Intern Med. 2002 Nov;252(5):389-97. doi: 10.1046/j.1365-2796.2002.01040.x. PMID 12528756
- [Background] Favus MJ, Karnauskas AJ, Parks JH, Coe FL. Peripheral blood monocyte vitamin D receptor levels are elevated in patients with idiopathic hypercalciuria. J Clin Endocrinol Metab. 2004 Oct;89(10):4937-43. doi: 10.1210/jc.2004-0412. PMID 15472188
- [Background] Frumar AM, Meldrum DR, Geola F, Shamonki IM, Tataryn IV, Deftos LJ, Judd HL. Relationship of fasting urinary calcium to circulating estrogen and body weight in postmenopausal women. J Clin Endocrinol Metab. 1980 Jan;50(1):70-5. doi: 10.1210/jcem-50-1-70. PMID 7350188
- [Background] Giannini S, Nobile M, Dalle Carbonare L, Lodetti MG, Sella S, Vittadello G, Minicuci N, Crepaldi G. Hypercalciuria is a common and important finding in postmenopausal women with osteoporosis. Eur J Endocrinol. 2003 Sep;149(3):209-13. doi: 10.1530/eje.0.1490209. PMID 12943523
- [Background] Lobo RA, Roy S, Shoupe D, Endres DB, Adams JS, Rude RK, Singer FR. Estrogen and progestin effects on urinary calcium and calciotropic hormones in surgically-induced postmenopausal women. Horm Metab Res. 1985 Jul;17(7):370-3. doi: 10.1055/s-2007-1013545. PMID 3161813
- [Background] McKane WR, Khosla S, Burritt MF, Kao PC, Wilson DM, Ory SJ, Riggs BL. Mechanism of renal calcium conservation with estrogen replacement therapy in women in early postmenopause--a clinical research center study. J Clin Endocrinol Metab. 1995 Dec;80(12):3458-64. doi: 10.1210/jcem.80.12.8530583.
- [Background] Nordin BE, Horowitz M, Need A, Morris HA. Renal leak of calcium in post-menopausal osteoporosis. Clin Endocrinol (Oxf). 1994 Jul;41(1):41-5. doi: 10.1111/j.1365-2265.1994.tb03782.x. PMID 8050130
- [Background] Nordin BE, WIshart JM, Clifton PM, McArthur R, Scopacasa F, Need AG, Morris HA, O'Loughlin PD, Horowitz M. A longitudinal study of bone-related biochemical changes at the menopause. Clin Endocrinol (Oxf). 2004 Jul;61(1):123-30. doi: 10.1111/j.1365-2265.2004.02066.x. PMID 15212654
- [Background] Nordin BE, Need AG, Morris HA, Horowitz M. Biochemical variables in pre- and postmenopausal women: reconciling the calcium and estrogen hypotheses. Osteoporos Int. 1999;9(4):351-7. doi: 10.1007/s001980050158. PMID 10550453
- [Background] Nordin BE, Need AG, Morris HA, Horowitz M, Robertson WG. Evidence for a renal calcium leak in postmenopausal women. J Clin Endocrinol Metab. 1991 Feb;72(2):401-7. doi: 10.1210/jcem-72-2-401. PMID 1991810
- [Background] Puche RC, Roveri E, Perez Jimeno N, Roberti A, Poudes G, Bocanera R, Tozzini R. Hypercalciuria and urinary saturation measurements in climacteric women. Maturitas. 1993 Jan;16(1):39-47. doi: 10.1016/0378-5122(93)90132-2. PMID 8429802
- [Background] Stock JL, Coderre JA, Mallette LE. Effects of a short course of estrogen on mineral metabolism in postmenopausal women. J Clin Endocrinol Metab. 1985 Oct;61(4):595-600. doi: 10.1210/jcem-61-4-595. PMID 2993339
- [Background] Voetberg GA, Netelenbos JC, Kenemans P, Peters-Muller ER, van de Weijer PH. Estrogen replacement therapy continuously combined with four different dosages of dydrogesterone: effect on calcium and lipid metabolism. J Clin Endocrinol Metab. 1994 Nov;79(5):1465-9. doi: 10.1210/jcem.79.5.7962344.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transdermal Estradiol
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study terminated. | 1

BASELINE CHARACTERISTICS:
Population: data were not collected
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0
Age, Continuous — Population: Study terminated
Sex: Female, Male — Population: Study terminated.
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in 24 Hour Urinary Calcium Excretion
Description: 0 participants were measured because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: 0 participants were analyzed because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

2. Secondary Outcome: Serum 1,25-dihydroxyvitamin D3
Description: 0 participants were analyzed because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: The study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

3. Secondary Outcome: Serum Bone Morphogenetic Protein 2
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

4. Secondary Outcome: Serum Sclerostin
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Serum Estradiol
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Serum Total Calcium
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Calculated Serum Ionized Calcium
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Calculated Tubular Resorption of Calcium
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Serum 25 Hydroxyvitamin D
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Serum Parathyroid Hormone
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Serum Phosphorus
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Serum Osteocalcin
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Serum Bone-specific Alkaline Phosphatase
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Serum C-telopeptides of Type 1 Collagen
Description: Not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Serum Procollagen Type 1 N-terminal Propeptide
Description: It is not available because the study was terminated
Time Frame: 4 weeks, 8 weeks
Population: Not available because the study was terminated
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The study was not finished and adverse events were not collected
Arm/Group | Transdermal Estradiol
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to 0 subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes